CLINICAL TRIAL: NCT05688241
Title: Epstein-Barr Virus (EBV) -Specific T Memory Stem Cell (Tscm) Therapy to Treat EBV- Driven Lymphomas/ Diseases
Brief Title: EBV-Tscm Cytotoxic T Cells (CTLs) for EBV- Driven Lymphomas/ Diseases
Acronym: ESPECT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01210; am22Khanna
Record Dates: First submitted 2022-12-21; First posted 2023-01-18 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: EBV Lymphoma; Post-transplant Lymphoproliferative Disease (PTLD)
Keywords: EBV-driven Lymphomas; EBV disease; Epstein-Barr Virus (EBV); Memory Stem Cell Therapy; Epstein-Barr Virus-specific T Memory Stem Cell Therapy (EBV-Tscm); cytotoxic T-cell line (CTL); T memory stem cells (Tscm); T-cell receptor (TCR); post-transplant lymphoproliferative disease (PTLD); Wnt-β-catenin inhibition; hematopoietic cell transplantation (HCT); Hematopoietic stem cell transplantation (HSCT)
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Intervention Model Description: Multi-center open-label, non-randomized phase I/II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: patients who undergo allogeneic HCT (Experimental): Patients with EBV driven lymphomas (e.g., natural killer (NK)/T-cell lymphoma), with EBV complications (e.g. haemophagocytic lymphohistiocytosis (HLH), CAEBV) or patients with primary immunodeficiency disorders with high risk for EBV complications (e.g. SCID) with planned allogeneic HCT.
  Interventions: Drug: Donor-derived ex-vivo expanded EBV Tscm CTL
- Group B: patients after HCT or SOT (Experimental): EBV-driven PTLD that develop after a HCT or solid organ transplantation (SOT) and show decreased response to rituximab.
  Interventions: Drug: Donor-derived ex-vivo expanded EBV Tscm CTL

INTERVENTIONS:
Drug: Donor-derived ex-vivo expanded EBV Tscm CTL — Cryopreserved cells will be thawed and infused at three time points. Dosing will be 2x10e6 EBV CTLs per kg of body weight. No prior lymphodepletion will be performed.

SUMMARY:
In this multi-center open-label, non-randomized phase I/II intervention study three consecutive doses of donor-derived EBV Tscm-CTLs will be administered to 10 patients with treatment-refractory EBV lymphoma, diseases or PTLDs. EBV Tscm-CTLs will derive from hematopoietic cell transplant (HCT) or third-party donors.

DETAILED DESCRIPTION:
Epstein Barr virus (EBV)-driven lymphomas and diseases are associated with poor prognosis. EBV proteins are recognized by T cells providing opportunities for EBV-specific T-cell therapy. Recent findings show that early differentiated T cells (T memory stem cells, Tscm) improve the prognosis in chronic viral diseases and are associated with effective tumor cell killing in melanoma patients. Tscm might be superior to highly differentiated T cells because of their longevity, robust proliferative potential, and capacity to reconstitute a wide T-cell receptor (TCR) diversity. This project will test the hypothesis that Tscm are efficacious for EBV-specific T-cell therapy. Clinical-grade enriched EBV-specific Tscm-CTLs will be prepared and used to treat patients with primary EBV lymphomas, diseases or post-transplant lymphoproliferative disease (PTLD) with limited other treatment options.

ELIGIBILITY:
Patients' inclusion criteria:

* Group A: Patients with EBV driven lymphomas (e.g., NK/T-cell lymphoma), with EBV complications (e.g. HLH, CAEBV) or patients with primary immunodeficiency disorders with high risk for EBV complications (e.g. SCID) with planned allogeneic HCT
* Group B: EBV-driven PTLD that develop after a HCT or SOT

For both groups:

* All age groups
* Negative pregnancy test in female patients of childbearing potential.
* Signed written informed consent of patient or/and parents

Patients' exclusion criteria:

* Patients receiving anti-thymocyte globulin or Campath within 28 days of infusion
* Patients with active, acute GvHD grades III-IV
* Previous severe reaction to dimethylsulfoxide (DMSO)

Donors' inclusion criteria:

* EBV positive serology (VCA and Epstein-Barr nuclear antigen (EBNA) immunoglobulin G (IgG) positive)
* Detectable interferon (IFN)-y-secreting T cells (>100 SFC/10e6 PBMC) measured by Elispot to the EBV consensus peptide pool
* Suitability for blood or HCT donation meeting requirements of local institutional guidelines
* An informed consent for EBV Tscm CTL manufacturing
* Age > 18 years

Donors' exclusion criteria:

* Detectable IFN-y-secreting T-cells <100 spot-forming cell (SFC)/10e6 PBMC measured by Elispot to EBV select
* Unwilling and/or unable to donate, according to the donor center

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of feasibility to expand Tscm-enriched EBV CTLs | one time assessment on day 9-11 of expansion before cryopreservation (plus at least 7 days for microbiological culture)
  Feasibility is defined as meeting the release criteria of EBV Tscm-CTL endproduct.
  Release criteria for the EBV Tscm-CTL follow Swissmedic Investigational Medicinal Product Dossier (IMPD). This includes viability of cluster of differentiation 3 (CD3)+ >70%, absolute CD3 count per kg of body weight per dose (≤2x10e6/kg), and a purity of CD3+ >90%. These criteria will be assessed before cryopreservation. A negative culture for bacteria and fungi for at least 7 days, endotoxin testing ≤5 EU/ml and negative result for Mycoplasma is required.
Safety of EBV Tscm-CTL infusion assessed by number of early infusion-related events | up to 12 hours after first dose of EBV Tscm-CTL infusion
  Number of early infusion-related events (early infusion-related events are clinically significant alterations of vital signs)
Safety of EBV Tscm-CTL infusion assessed by number of late clinical reaction to EBV Tscm-CTLs | from 12 hours after first dose until 3 months after the last dose of EBV CTLs
  Late clinical reaction to EBV Tscm-CTLs are signs of acute graft-versus-host disease (GvHD). Acute GVHD will be graded according to the modified Glucksberg criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Khanna, Prof. Dr. med., Principal Investigator — Klinik für Infektiologie und Spitalhygiene, University Hospital of Basel
Locations (8):
- Switzerland (8):
  - University Hospital Basel, Klinik für Infektiologie und Spitalhygiene, Basel
  - Universitäts-Kinderspital beider Basel (UKBB), Basel
  - Universitätsspital Bern, Klinik für Infektiologie, Bern
  - Hôpitaux Universitaires de Genève, Hôpital des Enfants, Geneva
  - Hôpitaux Universitaires de Genève, Service d'Hématologie, Geneva
  - Centre hospitalier universitaire vaudois, Service et Laboratoire central d'hématologie, Lausanne
  - Kinderspital Zürich, Zurich
  - University Hospital Zurich, Hämatologie, Zurich